CLINICAL TRIAL: NCT01657370
Title: A Phase IIb, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Pharmacokinetic Study of MK-1602 in the Treatment of Acute Migraine
Brief Title: A Pharmacokinetic Study of MK-1602 in the Treatment of Acute Migraine (MK-1602-007)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1602-007
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Results first posted 2016-12-09 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-10

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — ubrogepant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Placebo (Placebo Comparator): MK-1602 placebo-matching tablet orally for 3 doses: Dose 1 at the onset of a moderate or severe migraine (Day 1), Dose 2 in the evening of Day 3 and Dose 3 on Day 4. After 2 hours participants were able to take rescue medication if necessary.
  Interventions: Drug: Placebo; Drug: Rescue medication
- MK-1602 1 mg (Experimental): MK-1602 1 mg tablet orally for 3 doses: Dose 1 at the onset of a moderate or severe migraine (Day 1), Dose 2 in the evening of Day 3 and Dose 3 on Day 4. After 2 hours participants were able to take rescue medication if necessary.
  Interventions: Drug: MK-1602; Drug: Rescue medication
- MK-1602 10 mg (Experimental): MK-1602 10 mg tablet orally for 3 doses: Dose 1 at the onset of a moderate or severe migraine (Day 1), Dose 2 in the evening of Day 3 and Dose 3 on Day 4. After 2 hours participants were able to take rescue medication if necessary.
  Interventions: Drug: MK-1602; Drug: Rescue medication
- MK-1602 25 mg (Experimental): MK-1602 25 mg tablet orally for 3 doses: Dose 1 at the onset of a moderate or severe migraine (Day 1), Dose 2 in the evening of Day 3 and Dose 3 on Day 4. After 2 hours participants were able to take rescue medication if necessary.
  Interventions: Drug: MK-1602; Drug: Rescue medication
- MK-1602 50 mg (Experimental): MK-1602 50 mg tablet orally for 3 doses: Dose 1 at the onset of a moderate or severe migraine (Day 1), Dose 2 in the evening of Day 3 and Dose 3 on Day 4. After 2 hours participants were able to take rescue medication if necessary.
  Interventions: Drug: MK-1602; Drug: Rescue medication
- MK-1602 100 mg (Experimental): MK-1602 100 mg tablet orally for 3 doses: Dose 1 at the onset of a moderate or severe migraine (Day 1), Dose 2 in the evening of Day 3 and Dose 3 on Day 4. After 2 hours participants were able to take rescue medication if necessary.
  Interventions: Drug: MK-1602; Drug: Rescue medication

INTERVENTIONS:
Drug: MK-1602 — Three administrations of the same dose of MK-1602 on separate days. All 3 doses are either 1, 10, 25, 50 or 100 mg of MK-1602. Dose 1: Taken at onset of migraine of moderate or severe intensity. Dose 2: Taken the evening before Visit 2. Dose 3: Taken at Visit 2, which is Day 4 post migraine treatment (Dose 1).
  Dosage form is film coated tablet for oral administration.
  Arms: MK-1602 1 mg; MK-1602 10 mg; MK-1602 100 mg; MK-1602 25 mg; MK-1602 50 mg
Drug: Placebo — Three administrations of placebo for MK-1602 on separate days. Dose 1: Taken at onset of migraine of moderate or severe intensity. Dose 2: Taken the evening before Visit 2. Dose 3: Taken at Visit 2, which is Day 4 post migraine treatment (Dose 1).
  Dosage form is film coated tablet for oral administration.
  Arms: Placebo
Drug: Rescue medication — If moderate or severe migraine headache pain continues 2 hours after dose of study medication or if migraine headache comes back within 48 hours,
  Participants will be allowed to take their own rescue migraine medication, which may include analgesics (e.g., nonsteroidal anti-inflammatory drugs [NSAIDs]), anti-emetics, triptans, opiates or other medication not explicitly excluded.

SUMMARY:
The purpose of this study is to characterize the pharmacokinetics of MK-1602 in the treatment of acute migraine, including the influence of demographic and other variables on MK-1602 pharmacokinetics, and to evaluate the relationship between MK-1602 concentrations and efficacy of the drug.

ELIGIBILITY:
Inclusion Criteria:

* > 1 year history of migraine with or without aura as defined by International Headache Society (IHS) criteria 1.1 and/or 1.2
* Migraines typically last between 4 to 72 hours, if untreated
* ≥ 2 and ≤ 8 moderate or severe migraine attacks per month in each of

the two months prior to screening

* Male, female who is not of reproductive potential, or female of

reproductive potential with a screening serum β-human chorionic gonadotropin (β-hCG) level consistent with a not-pregnant state, and who agrees to use acceptable contraception

Exclusion Criteria:

* Pregnant or breast-feeding, or is a female expecting to conceive within the projected duration of study participation
* Participant has difficulty distinguishing his/her migraine attacks from tension-type headaches
* History of predominantly mild migraine attacks or migraines that usually

resolve spontaneously in less than two hours

* More than 15 headache-days per month or has taken medication for acute headache on more than 10 days per month in any of the three months prior to screening
* Basilar-type or hemiplegic migraine headache
* > 50 years old at age of migraine onset
* Taking migraine prophylactic medication where the prescribed daily dose

has changed during the 3 months prior to screening and during the study

* Taking a proton pump inhibitor (PPI) or a histamine receptor 2 (H2) blocker on a daily or near daily basis (> 3 days per week)
* Taking the following medications from 1 month prior to screening through study period: potent cytochrome P450 (CYP) 3A4 inhibitors (e.g., cyclosporine, itraconazole, ketoconazole, fluconazole, erythromycin, clarithromycin, nefazodone, telithromycin, cimetidine, quinine, diltiazem, verapamil, modafinil and human immunodeficiency virus [HIV] protease inhibitors), moderate or marked CYP3A4 inducers (e.g., rifampicin, rifabutin, barbiturates [e.g., phenobarbital and primidone], systemic glucocorticoids, nevirapine, efavirenz, pioglitazone, carbamazepine, phenytoin, and St. Johns wort), or drugs with narrow therapeutic margins and potential for drug interactions in the CYP2C family (e.g., warfarin)
* Participant is unable to refrain from consumption of grapefruit or grapefruit juice during study
* History of hypersensitivity to, or has experienced a serious adverse event

in response to 3 or more classes of drugs (prescription and over-the-counter)

* Clinical or laboratory evidence of uncontrolled diabetes, HIV disease, or significant pulmonary, renal, hepatic, endocrine, or other systemic disease
* Other confounding pain syndromes, psychiatric conditions such as uncontrolled major depression, dementia or significant neurological disorders other than migraine. Patients who are currently being treated with non-prohibited medication for depression and symptoms are well controlled are eligible to participate
* Participant is at imminent risk of self-harm
* History of malignancy ≤ 5 years prior to study, except for adequately treated basal cell or squamous cell skin cancer, or in situ cervical cancer
* History of gastric or small intestinal surgery (including gastric bypass

surgery or banding), or presence of a disease that causes malabsorption

* History or current evidence of any condition, therapy, lab abnormality or

other circumstance that might confound the results of the study, or interfere with subject's participation for the full duration of the study

* Participant has recent history (within the last year) of drug or alcohol abuse or dependence or is a user of recreational or illicit drugs
* Participant is legally or mentally incapacitated
* Donation of blood products or phlebotomy of > 300 ml within 8

weeks of study, or intent to donate blood products or receive

blood products within 30 days of screening and throughout study

* Intent to donate eggs or sperm within the projected duration of the

study

* Current participation in or participation within 30 days of screening

in a study with an investigational compound or device, with the exception of MK-1602 Protocol 006

* Previous exposure to MK-0974 and/or MK-3207
* Use within the past 2 months of an opioid- or barbiturate-containing

analgesic for migraine relief

* Inpatient or emergency department treatment of an acute migraine

attack within the past 2 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195 (Actual)
Dates: Start 2012-08; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Started | 33 | 32 | 32 | 33 | 34 | 31
Completed | 27 | 28 | 25 | 28 | 27 | 27
Not Completed | 6 | 4 | 7 | 5 | 7 | 4
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0 | 1
Not completed — Physician Decision | 2 | 3 | 1 | 2 | 5 | 0
Not completed — Lack of Qualifying Event | 1 | 0 | 3 | 2 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 1 | 1 | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 0 | 1 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All Subjects as Treated Population included all randomized participants who received at least 1 dose of study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg | Total
Number analyzed (Participants) | 28 | 28 | 26 | 28 | 28 | 27 | 165
Age, Customized [Number; unit: participants]
  <20 years | 1 | 1 | 0 | 0 | 0 | 2 | 4
  20 to 29 years | 4 | 8 | 6 | 9 | 11 | 9 | 47
  30 to 39 years | 9 | 7 | 7 | 7 | 6 | 6 | 42
  40 to 49 years | 9 | 9 | 7 | 7 | 6 | 6 | 44
  50 to 59 years | 5 | 3 | 4 | 3 | 4 | 3 | 22
  60 to 64 years | 0 | 0 | 0 | 2 | 0 | 1 | 3
  >= 65 years | 0 | 0 | 2 | 0 | 1 | 0 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 22 | 23 | 26 | 18 | 140
  Male | 3 | 2 | 4 | 5 | 2 | 9 | 25

OUTCOME MEASURES:

1. Primary Outcome: Dry Blood Spot (DBS) MK-1602 Concentration at 2 Hours Post-Dose on Migraine Treatment Day
Description: The participant collected blood by fingerstick on a card. The card was sent to a laboratory and the concentration of MK-1602 determined using the dried blood spot (DBS) assay.
Time Frame: 2 hours post dose 1
Population: Participants from the Pharmacokinetic Analysis Population, all participant who received treatment, with data available for analysis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanomolar (nM)
Arm/Group | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 21 | 23 | 27 | 22 | 23
nanomolar (nM) | 1.9 (73) | 17.0 (74) | 43.8 (130) | 52.7 (270) | 184.8 (170)

2. Primary Outcome: Percentage of Participants Reporting Pain Freedom (PF) at 2 Hours Post-Dose on Migraine Treatment Day
Description: PF was defined as a decrease from a moderate or severe migraine headache (Grade 2 or 3) at Baseline to no pain (Grade 0) 2 hours post-dose. Headache severity was reported by the participant using a 4-point scale where: 0=no pain, 1=mild pain, 2=moderate pain and 3=severe pain.
Time Frame: 2 hours post dose 1
Population: Full Analysis Set included all participants who received study treatment, had a Baseline headache severity measurement, and at least one post-dose efficacy measurement prior to, or including, the 2-hour time point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 28 | 28 | 26 | 28 | 28 | 27
percentage of participants | 0.0 [0.0 to 12.3] | 0.0 [0.0 to 12.3] | 3.8 [0.1 to 19.6] | 17.9 [6.1 to 36.9] | 28.6 [13.2 to 48.7] | 11.1 [2.4 to 29.2]

3. Primary Outcome: Percentage of Participants With Pain Relief (PR) at 2 Hours Post-Dose on Migraine Treatment Day
Description: PR was defined as a decrease from a moderate or severe migraine headache (Grade 2 or 3) at Baseline to a mild headache or no headache (Grade 1 or 0) 2 hours post dose. Headache severity was reported by the participant using a 4-point scale where: 0=no pain, 1=mild pain, 2=moderate pain and 3=severe pain.
Time Frame: 2 hours post dose 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 28 | 28 | 26 | 28 | 28 | 27
percentage of participants | 42.9 [24.5 to 62.8] | 42.9 [24.5 to 62.8] | 30.8 [14.3 to 51.8] | 46.4 [27.5 to 66.1] | 67.9 [47.6 to 84.1] | 70.4 [49.8 to 86.2]

4. Secondary Outcome: Percentage of Participants Reporting Absence of Phonophobia at 2 Hours Post-Dose on Migraine Treatment Day
Description: Phonophobia is sensitivity to sound.
Time Frame: 2 hours post dose 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 28 | 28 | 26 | 28 | 28 | 27
percentage of participants | 28.6 [13.2 to 48.7] | 42.9 [24.5 to 62.8] | 30.8 [14.3 to 51.8] | 42.9 [24.5 to 62.8] | 57.1 [37.2 to 75.5] | 44.4 [25.5 to 64.7]

5. Secondary Outcome: Percentage of Participants Reporting Absence of Photophobia at 2 Hours Post-Dose on Migraine Treatment Day
Description: Photophobia is sensitivity to light.
Time Frame: 2 hours post dose 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 28 | 28 | 26 | 28 | 28 | 27
percentage of participants | 25.0 [10.7 to 44.9] | 25.0 [10.7 to 44.9] | 26.9 [11.6 to 47.8] | 28.6 [13.2 to 48.7] | 46.4 [27.5 to 66.1] | 48.1 [28.7 to 68.1]

6. Secondary Outcome: Percentage of Participants Reporting Absence of Nausea at 2 Hours Post-Dose on Migraine Treatment Day
Time Frame: 2 hours post dose 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 28 | 28 | 26 | 28 | 28 | 27
percentage of participants | 67.9 [47.6 to 84.1] | 57.1 [37.2 to 75.5] | 69.2 [48.2 to 85.7] | 57.1 [37.2 to 75.5] | 82.1 [63.1 to 93.9] | 74.1 [53.7 to 88.9]

7. Secondary Outcome: Percentage of Participants With Sustained Pain Freedom (SPF) From 2-24 Hours Post-Dose on Migraine Treatment Day
Description: SPF was defined as PF at 2 hours post-dose, with no administration of any rescue medication and with no occurrence of a mild/moderate/severe headache during the 2-24 hour period after dosing with study medication.
Time Frame: 2-24 hours post dose 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 28 | 28 | 26 | 28 | 28 | 27
percentage of participants | 0.0 [0.0 to 12.3] | 0.0 [0.0 to 12.3] | 3.8 [0.1 to 19.6] | 10.7 [2.3 to 28.2] | 14.3 [4.0 to 32.7] | 3.7 [0.1 to 19.0]

8. Secondary Outcome: Percentage of Participants With Sustained Pain Relief (SPR) From 2-24 Hours Post-Dose on Migraine Treatment Day
Description: SPR was defined as PR at 2 hours post-dose, with no administration of any rescue medication and with no occurrence of a moderate/severe headache during the 2-24 hour period after dosing with study medication.
Time Frame: 2-24 hours post dose 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 28 | 28 | 26 | 28 | 28 | 27
percentage of participants | 28.6 [13.2 to 48.7] | 25.0 [10.7 to 44.9] | 15.4 [4.4 to 34.9] | 42.9 [24.5 to 62.8] | 57.1 [37.2 to 75.5] | 48.1 [28.7 to 68.1]

9. Secondary Outcome: Percentage of Participants With Total Migraine Freedom (TMF) at 2 Hours Post-Dose on Migraine Treatment Day
Description: TMF at 2 hours post-dose was defined as PF with no photophobia, phonophobia, nausea, or vomiting at 2 hours post-dose.
Time Frame: 2 hours post dose 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 28 | 28 | 26 | 28 | 28 | 27
percentage of participants | 0.0 [0.0 to 12.3] | 0.0 [0.0 to 12.3] | 0.0 [0.0 to 13.2] | 14.3 [4.0 to 32.7] | 28.6 [13.2 to 48.7] | 7.4 [0.9 to 24.3]

10. Secondary Outcome: Percentage of Participants With TMF From 2-24 Hours Post-Dose on Migraine Treatment Day
Description: TMF from 2-24 hours post-dose was defined as SPF with no photophobia, phonophobia, nausea, or vomiting during the 2-24 hour period after dosing with study medication.
Time Frame: 2-24 hours post dose 1
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 28 | 28 | 26 | 28 | 28 | 27
percentage of participants | 0.0 [0.0 to 12.3] | 0.0 [0.0 to 12.3] | 0.0 [0.0 to 13.2] | 10.7 [2.3 to 28.2] | 14.3 [4.0 to 32.7] | 3.7 [0.1 to 19.0]

11. Other Pre Specified Outcome: Dry Blood Spot (DBS) MK-1602 Concentrations on Migraine Treatment Day
Time Frame: Up to 24 hours post dose 1
Population: As per protocol, only listings of individual DBS for MK-1602 over time were produced. No formal non-compartmental Pharmacokinetic (PK) analysis was done for this outcome measure.
Arm/Group | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

12. Other Pre Specified Outcome: Dry Blood Spot MK-1602 Concentration at 3.5 Hours Post-Dose at Visit 2 (Day 4)
Time Frame: 3.5 hours post dose 3
Population: As per protocol, only listings of individual DBS concentrations for MK-1602 over time were produced. No formal non-compartmental PK analysis was done for this outcome measure.
Arm/Group | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

13. Other Pre Specified Outcome: Plasma MK-1602 Concentrations at Visit 2 (Day 4)
Time Frame: Up to 3.5 hours post dose 3
Population: As per protocol, only listings of individual plasma concentrations for MK-1602 over time were produced. No formal non-compartmental PK analysis was done for this outcome measure.
Arm/Group | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: All Subjects as Treated Population, all randomized participants who received at least 1 dose of study treatment, was used to determine the number of participants at risk for Serious Adverse Events and Other Adverse Events.
Arm/Group | Placebo | MK-1602 1 mg | MK-1602 10 mg | MK-1602 25 mg | MK-1602 50 mg | MK-1602 100 mg
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/28 | 0/26 | 0/28 | 0/28 | 0/27
Other Adverse Events (participants affected / at risk) | 6/28 | 6/28 | 2/26 | 10/28 | 7/28 | 7/27
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=28) | MK-1602 1 mg (N=28) | MK-1602 10 mg (N=26) | MK-1602 25 mg (N=28) | MK-1602 50 mg (N=28) | MK-1602 100 mg (N=27)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 2 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 2 | 1
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 2 | 3 | 1
Fatigue (General disorders) | 1 | 0 | 0 | 2 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 0 | 1 | 0 | 2
Dizziness (Nervous system disorders) | 4 | 2 | 0 | 2 | 0 | 2
Headache (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.